CLINICAL TRIAL: NCT03659201
Title: Randomized Clinical Trial, Placebo Controlled and Active Comparator, to Evaluate Efficacy and Safety of Neosil in Chronic Effluvium
Brief Title: Efficacy and Safety of Neosil on Chronic Effluvium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMS (Industry)
Collaborators: Luxbiotech (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAEP 0100118PC - Si+Biobetter
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Chronic Telogen Effluvium
MeSH Terms: interventions — pantogar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neosil complete (Experimental): The patient will take the tablets, as follow:
  3 tablets of Neosil, Oral, per day - during the initial 12 weeks; and
  2 tablets of Neosil Oral, per day - during the last 12 weeks.
  Interventions: Drug: Neosil complete
- Pantogar (Experimental): The patient wil take the tablets, as follow:
  3 tablets of Placebo, Oral, per day - during the initial 12 weeks; and
  3 tablets of Pantogar, Oral, per day - during the last 12 weeks.
  Interventions: Drug: Pantogar
- Neosil (Experimental): The patient will take the tablets, as follow:
  2 tablets of Neosil Oral, per day - during the 12 weeks.
  Interventions: Drug: Neosil

INTERVENTIONS:
Drug: Neosil complete — Oral, during 24 weeks.
  Arms: Neosil complete
Drug: Pantogar — Oral, placebo for 12 weeks and pantogar for 12 weeks.
  Arms: Pantogar
Drug: Neosil — Oral, during only 12 weeks.
  Arms: Neosil

SUMMARY:
The purpose of this study is to evaluate the efficacy of Neosil in the treatment of chronic effluvium

ELIGIBILITY:
Inclusion Criteria:

* Participants who present hair loss for more than 6 months;
* Do not use other possible cosmetic or dermatological treatments, during the trial;
* Not change the diet during the trial and not be any restrictive diet during this period.

Exclusion Criteria:

* Pregnancy or risk of pregnancy and lactating patients;
* Use of any products to promote hair growth within the 6 months prior to the Baseline Visit;
* History of hair transplants;
* Current skin disease;
* History hypersensitivity to the active ingredients used in the study;
* Participation in clinical trial in the year prior to this study;
* Known history of non controled systemic disease (diabetes, hypertension, anemia, iron deficiency, and others);
* Gastric diseases;
* Smoker;
* History of systemic disease (HIV, non specify autoimmune disease, hepatitis, and others).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Hair density | 24 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Caep Centro Avancado de Estudos E Pesquisas Ltda, Campinas, São Paulo, Brazil